CLINICAL TRIAL: NCT06858891
Title: The Effect of Transversus Abdominis Plane Block on Maternal-Infant Bonding in Cesarean Sections Performed Under Spinal Anesthesia
Brief Title: The Effect of TAP Block on Maternal-Infant Bonding
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Nezir Yılmaz, Associate Professor, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: ADYU-NYILMAZ--007
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Cesarean Section; Transversus Abdominis Plane (TAP) Block
Keywords: cesarean section; Transversus Abdominis Plane (TAP) Block; Maternal-Infant Bonding
MeSH Terms: conditions — Bites and Stings | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two groups using the sealed-envelope method: one group will receive bilateral transversus abdominis plane (TAP) block in addition to standard care, while the other group will receive only standard pain management.
Who Masked: Investigator
Masking Description: The researchers performing the block procedures were not involved in the postoperative assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): standard pain management
- Block group (Experimental): standard pain management + Bilateral TAP block
  Interventions: Procedure: Transversus abdominis plane (TAP) block

INTERVENTIONS:
Procedure: Transversus abdominis plane (TAP) block — Under ultrasound guidance, 20 cc of 0.25% bupivacaine was planned to be administered between the internal oblique and transversus abdominis fascial planes on both lateral aspects of the anterior abdominal wall.
  Arms: Block group

SUMMARY:
Cesarean delivery is a common surgical procedure that is typically performed under spinal anesthesia. Postoperative pain management has a significant impact on both the mother's physical recovery and the quality of maternal-infant bonding. The quality of maternal-infant bonding is influenced by various factors, including postoperative pain, early mobilization, initiation of breastfeeding, stress, psychological status, and hormonal balance. Studies have reported that adequate postoperative pain management, early breastfeeding, and early mobilization have positive effects on maternal-infant bonding.

Transversus abdominis plane (TAP) block is a regional anesthesia technique known for its efficacy in controlling postoperative pain. Bilateral TAP block performed after cesarean section has been associated with lower pain scores, reduced analgesic consumption, and shorter hospital stays. However, its impact on maternal-infant bonding has not been fully elucidated.

This study aims to investigate the effect of bilateral TAP block on maternal-infant bonding in women undergoing cesarean section under spinal anesthesia.

DETAILED DESCRIPTION:
This study aims to investigate the effect of TAP block on maternal-infant bonding in women undergoing cesarean section under spinal anesthesia. Participants will be randomly assigned to two groups: one group will receive a TAP block in addition to standard care, while the other group will receive only standard pain management. Maternal-infant bonding will be assessed using the maternal bonding scale and behavioral evaluations at 48 hours and one month postpartum.

The primary outcome is to evaluate whether the TAP block improves early bonding by reducing pain and enhancing maternal comfort. Secondary outcomes include maternal pain scores, mobilization time, and initiation of breastfeeding. This study aims to contribute to the optimization of pain management strategies in cesarean deliveries, ultimately improving both maternal recovery and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 aged or older patients,
* Agree to participate in the study
* Pregnant women without any maternal or fetal pathology during the pregnancy.

Exclusion Criteria:

* <18 age
* Deny to participate in the study
* maternal or fetal pathology during the pregnancy
* Allergy to local anesthetics
* local ingection at block side

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cesarean Section
Enrollment: 132 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-04-05 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Perceived Maternal Parenting Self-Efficacy (PMP S-E) score | Postoperative 48th hour, based on a single assessment
  The PMP S-E is a questionnaire consisting of 18 questions that assess the mother's bond with her baby and her sense of parenthood. Each question consists of 4 options and will be scored on a scale from 0 to 3. The total score of the questionnaire will range from 0 to 54.

SECONDARY OUTCOMES:
Visual Analog scale (VAS) score | Postoperative 2th, 4th, 6th, 12th and 24th hours
  Postoperative pain scores will be assesed with visual analog scale at postoperative period. Vas score will range to 0-10. O refers to no pain and 10 refers to the worst pain ever had.

IPD SHARING:
Plan to Share IPD: Undecided